CLINICAL TRIAL: NCT07121582
Title: Modulation of Beta Oscillatory Rhythms in Stroke to Promote Corticomuscular Circuit Function
Brief Title: Modulation of Brain Rhythms in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 25-1318; 1R21HD117319 (NIH)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: stroke; neurostimulation; brain; motor; hand; electroencephalography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a randomized, two-sequence (AB I BA), two-treatment crossover study design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor then Visual Brain Stimulation (Experimental): Following the first block of 20 grip/squeeze trials completed without brain stimulation, participants will complete a second and third set of blocks where non-invasive brain stimulation just before each grip trial will occur. Participants randomized to the "motor then visual brain stimulation" arm will receive stimulation to the motor part of their brain first followed by non-invasive brain stimulation to the visual (occipital) part of the brain. A 10-15 min participant break will separate the delivery of motor and visual brain stimulation (i.e., second and third blocks).
  Interventions: Other: Motor Brain Stimulation; Other: Visual Brain Stimulation
- Visual then Motor Brain Stimulation (Experimental): Following the first block of 20 grip/squeeze trials completed without brain stimulation, participants will complete a second and third set of blocks where non-invasive brain stimulation just before each grip trial will occur. Participants randomized to the "visual then motor brain stimulation" arm will receive stimulation to the visual part of their brain first followed by non-invasive brain stimulation to the motor part of the brain. A 10-15 min participant break will separate the delivery of visual and motor brain stimulation (i.e., second and third blocks).
  Interventions: Other: Motor Brain Stimulation; Other: Visual Brain Stimulation

INTERVENTIONS:
Other: Motor Brain Stimulation — For each grip trial (20 grip trials per block), participants will receive visual cues that signify the onset and offset of squeezing. Just prior to the start of the visual cue representing the onset of squeezing, participants will receive a burst of repetitive transcranial magnetic stimulation (rTMS) to their primary motor hotspot region. Motor brain stimulation will involve 3 bursts of 5 pulses/burst with a 20 Hz inter-pulse interval delivered at 90% of their resting or active motor threshold.
Other: Visual Brain Stimulation — For each grip trial (20 grip trials per block), participants will receive visual cues that signify the onset and offset of squeezing. Just prior to the start of the visual cue representing the onset of squeezing, participants will receive a burst of repetitive transcranial magnetic stimulation (rTMS) to their ipsilesional occipital cortex region. Visual brain stimulation will involve 3 burst of 5 pulses/burst with a 20 Hz inter-pulse interval delivered at 90% of their resting or active motor threshold.
  Other Names: Active Control Site; Decoy Site

SUMMARY:
The goal of this research study is to examine communication between brain and muscle in individuals with stroke and determine if applying non-invasive brain stimulation to different parts of the brain improves this communication and performance on a hand squeezing task.

The investigators will fit participants with an electroencephalography (EEG) cap and place electromyography (EMG) stickers on participants hand and arm muscles to record brain and muscle activity, respectively.

Participants will complete a single research visit lasting approximately 3 hours. During this visit, participants will receive two different types of non-invasive brain stimulation: [1] stimulation to the motor part of the brain and [2] stimulation to the visual part of the brain. Participants will be randomized so that half will receive stimulation to the motor part of the brain first followed by stimulation to the visual part of the brain second and vice versa. Participants will complete three blocks of hand squeezing trials using the stroke-affected (weak) hand. During the first block of squeezing trials, no brain stimulation will occur. During the second and third blocks, participants will receive stimulation just before each hand squeezing trial. The investigators will record participants' brain and muscle activity during these blocks of hand squeezing trials. Additionally, participants will also complete screening tests and exams looking at mood, motor function, and cognition.

DETAILED DESCRIPTION:
The purpose of this pilot study is to investigate and modulate corticomuscular coherence (CMC) by using beta-burst repetitive transcranial magnetic stimulation (rTMS). The central hypothesis is that the enhancement of neural oscillatory rhythms in the beta frequency range (13-30 Hz), which supports corticomuscular circuit function, will strengthen CMC measurement. Prior research has indicated that CMC, a surrogate measure of functional connectivity between the brain and peripheral muscles, has clinical relevance as a potential biomarker for motor recovery following stroke. In this cross-over study, the investigators will enroll 20 participants with chronic (≥ 6 months) stroke to complete a single research visit. The investigator will examine corticomuscular circuit function in response to beta-burst repetitive transcranial magnetic stimulation (rTMS) delivery to either participants' ipsilesional motor hotspot (active site) or ipsilesional occipital cortex (control site). The sequence or order of brain stimulation to the active and control site will be randomized across participants (described further below).

Participants will perform three blocks of a precision grip task with their stroke-affected (weak) hand using a custom-built dynamometer device. Each block will contain 20 trials for a total of 60 trials. Participants will receive visual cues when to squeeze the dynamometer device and when to relax their hand. They will also receive visual feedback of their force output to a visual target, which corresponds to 20% of their maximum voluntary contraction force. Prior to the start of these three blocks, participants will be randomized to a rTMS sequence (AB or BA). The first block of 20 trials does not involve stimulation delivery. Participants randomized to the AB sequence will receive rTMS stimulation to a "decoy" or active control site (ipsilesional occipital cortex) during the second block of 20 trials followed by stimulation to the active site (ipsilesional motor hotspot around primary motor cortex, M1) during the third block of 20 trials. Those randomized to the BA sequence will start with stimulation to the active site (M1) during the second block followed by stimulation to the ipsilesional occipital cortex during the third block. Stimulation will occur as a "burst" delivered just prior to the start of each grip trial that is the time just before participant's receive the visual cue to initiate the squeeze.

The investigators will also determine how the degree of injury to the ipsilesional corticospinal tract impacts responsively to beta-burst rTMS. The investigators will assess corticospinal excitability using single transcranial magnetic stimulation pulses to measure the downstream motor-evoked potential (MEP) response. Lastly, investigators will also determine if beta-burst rTMS impacts motor performance as assessed by reaction time and grip precision. The hypotheses are as follows:

1. greater pre/post change in CMC following beta-burst rTMS to the active brain site (M1/motor hotspot region) compared to the active control site (ipsilesional occipital cortex)
2. those with greater corticospinal tract injury, as denoted by reduced MEP amplitude and increased MEP latency, will demonstrate less pre-post change in CMC
3. beta-burst rTMS to the active site (M1/motor hotspot region) will result in improved grip task performance based on reduced reaction times and improved grip precision in comparison rTMS delivery to the ipsilesional occipital cortex (active control site).

ELIGIBILITY:
Inclusion Criteria:

* One and only one chronic (≥ 6 months) unilateral cortical/subcortical ischemic or hemorrhagic stroke as confirmed by medical records
* Upper extremity weakness (hemiparesis) contralateral to the stroke
* Sufficient cognitive capacity (Montreal Cognitive Assessment ≥ 26 points), communication function, and English proficiency to understand and safely comply with all study procedures
* Ipsilesional motor-evoked potential response
* Able to perform isometric grip task by making a fist with their stroke-affected hand (hand contralateral to the stroke)

Exclusion Criteria:

* Contraindications to TMS (seizure activity within past 2 years, pregnancy, indwelling metal)
* Cognitive deficits (Montreal Cognitive Assessment < 26 points)
* Concurrent physical/occupational therapy and/or clinical trial participation
* Injury or conditions that impact affected extremity-use beyond stroke (e.g., arthritis)
* Impaired vision despite use of aid (e.g. glasses, contacts, etc.)
* Cerebellar stroke
* Major medical/neurological/psychiatric condition impacting physical function in the opinion of the physician co-investigator
* Absent ipsilesional motor-evoked potential response

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Corticomuscular Coherence Change | Immediately (within 5 minutes) before and after (within 5 minutes) each stimulation block.
  Investigators will compute pre/post changes in brain-muscle functional connectivity (i.e., corticomuscular coherence, CMC) following across each block (20 trials/block). Specifically, investigators are focused on CMC in the beta (13-30 Hz) frequency range between the ipsilesional motor cortex (M1) and the affected first dorsal interossei muscle. Investigators will calculate CMC at two distinct phases during the squeezing task that correspond to the ramp/recruitment phase (i.e., squeezing to the target) and the hold/sustain phase (when participant's reach the target and sustain their grip).
Grip Precision | Immediately (within 5 minutes) before and after (within 5 minutes) each stimulation block.
  The variance of participants' force output from a visual target
Reaction Time | Immediately (within 5 minutes) before and after (within 5 minutes) each stimulation block.
  The time delay between the grip signal onset (visual cue provided to participants) and the realized force.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Cassidy, DPT, PT, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bondurant Hall, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that support the results will be shared. Data will include: Corticomuscular Coherence Measures, Behavioral Tests/Measures, motor-evoked potential data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared no later than 6 months after publication submission with no end date.
Access Criteria: Approved Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)'s Data and Specimen Hub (DASH).
URL: https://dash.nichd.nih.gov